CLINICAL TRIAL: NCT07024498
Title: Coordinating Outpatient bupreNorphiNe for Emergency Care and Continuing Treatment
Acronym: CONNECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2284130; R61DA059027 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
Keywords: emergency department; opioid use disorder; care coordination; implementation science; hybrid effectiveness-implementation; multiteam systems; buprenorphine; stepped wedge
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge design with intervention assignment at the site level and the primary outcome assessed at the patient level. The intervention will be implemented sequentially at the site level. The sequence in which sites will implement the intervention was determined prospectively to alternate between sites that did versus did not participate in the prior study to identify implementation strategies. After a 9 month baseline period, one site will transition to the intervention condition every 3 months until all four have implemented the intervention. Patients will be followed for up to 12 months after their ED visit to assess buprenorphine treatment outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospital ED and 2 associated outpatient clinics that provide buprenorphine treatment (Other): Each arm will receive the intervention at a different time point and will provide data for both the pre- and post-intervention conditions. During the pre-intervention periods, ED teams will use their existing workflows/procedures for referring patients to and coordinating with outpatient clinics that provide buprenorphine. During the post-implementation period, the ED and outpatient teams will use workflows/procedures that have incorporated the intervention.
  Interventions: Other: care coordination implementation strategies

INTERVENTIONS:
Other: care coordination implementation strategies — The intervention will be a bundle of implementation strategies developed during a prior study and informed by the multi-team systems framework. Core implementation strategies are expected to include a standardized ED substance use navigator note (with education and billing support), a mechanism for sharing PHI information across ED-clinic pairs that use different electronic health record systems, an improved ability for patients to directly contact EDs and clinics, ensuring ED and outpatient teams mutually understand each other roles, implementing procedures to increase capacity for same-day outpatient buprenorphine refills, and interactive problem solving with an external facilitation team. Strategies will be adapted to local contexts at each site.

SUMMARY:
The main purpose of this stepped wedge trial will be to test the impact of a bundle of implementation strategies designed to improve ED-outpatient care coordination on long-term buprenorphine retention among adult patients who start buprenorphine for opioid use disorder in a hospital emergency department (ED) and then are referred for continued outpatient buprenorphine treatment after they leave the ED. Our hypothesis is that adopting the bundle of implementation strategies will be associated with subsequent increases in:

A) Cumulative number of days with active buprenorphine prescription at 3, 6, and 12 months after patients' initial ED visit (6 months = primary outcome)

B) Proportion of patients with active buprenorphine prescriptions without gaps in buprenorphine coverage of more than 7 days at 3, 6, and 12 months after patients' initial ED visit

C) Proportion of patients who fill at least 1 outpatient buprenorphine prescription within 30 days of their ED visit

D) Clinician reported quality of ED-outpatient care coordination and care transitions

DETAILED DESCRIPTION:
Buprenorphine is a highly effective but underused medication for opioid use disorder that reduces cravings and decreases overdose risk. Starting buprenorphine for opioid use disorder in emergency departments (EDs) is recognized as a best clinical practice in the US. However, effective strategies to help patients sustain buprenorphine treatment after they leave the ED are urgently needed. To increase access to buprenorphine treatment, California established California Bridge, a state-funded program that offers same-day buprenorphine initiation plus referral to outpatient opioid use disorder treatment for patients. However, suboptimal ED-outpatient care coordination is a common barrier to buprenorphine retention. During a prior study, we identified a bundle of implementation strategies designed to improve ED-outpatient care coordination for patients who start buprenorphine for opioid use disorder in the ED. In this hybrid effectiveness-implementation study, the research team will work with core clinical teams at 12 sites (4 EDs and 8 outpatient clinics [2 clinics per ED]) to implement a bundle of implementation strategies at each site. Implementation will occur over a 12 month period (~3 months per site). Patient cohorts will be identified through electronic health record query reports. Data from eligible patients will then be abstracted from the electronic health record at each hospital. Changes in care coordination will be assessed using clinician surveys. Treatment outcomes will be assessed using buprenorphine prescription records obtained from California's prescription drug monitoring program linked to electronic health record data at the patient level. Study results will be used to develop an implementation blueprint that hospitals in California and across the US can use to improve opioid use disorder treatment outcomes for patients who start buprenorphine in hospital EDs.

ELIGIBILITY:
Inclusion Criteria:

* patients who start buprenorphine for opioid use disorder at a participating ED

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3492 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
buprenorphine treatment (continuous) | 6 months
  Cumulative number of days with active buprenorphine prescription after initial ED visit

SECONDARY OUTCOMES:
buprenorphine treatment (continuous) | 3 months, 12 months
  Cumulative number of days with active buprenorphine prescription after initial ED visit
buprenorphine retention (binary) | 3 months, 6 months, 12 months
  Proportion of patients with active buprenorphine prescriptions after initial ED visit without a gap in buprenorphine coverage of more than 7 days
outpatient buprenorphine initiation | 30 days
  Proportion of patients who fill at least 1 outpatient buprenorphine prescription within 30 days of their ED visit

OTHER OUTCOMES:
quality of care transitions | approximately 3 months after the implementation period at each site, controlling for baseline values
  Handoffs and transitions subscale of AHRQ Survey on Patient Safety Culture
quality of care coordination | approximately 3 months after the implementation period at each site, controlling for baseline values
  Teamwork across units subscale of AHRQ Survey on Patient Safety Culture

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Henry, MD MSc, Principal Investigator — University of California, Davis; Aimee K Moulin, MD MAS, Principal Investigator — University of California, Davis
Locations (4):
- United States (4):
  - El Centro Regional Medical Center Emergency Department, El Centro, California
  - University of California Irvine Emergency Department, Irvine, California
  - Marshall Medical Center Emergency Department, Placerville, California
  - University of California Davis Emergency Department, Sacramento, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be deposited in a public data registry as required by NIH HEAL data sharing guideilnes. However, due to state-level restrictions, individual level buprenorphine prescription data will not be shared.
Time Frame: expected 12 months after study completion